CLINICAL TRIAL: NCT00791947
Title: A Nordic Phase II Study of Peripheral T-cell Lymphomas Based on Dose-intensive Induction and High-dose Consolidation With Autologous Stem Cell Rescue
Brief Title: A Nordic Phase II Study of PTCL Based on Dose-intensive Induction and High-dose Consolidation With ASCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG-T-01; 2006-000389-35 (EudraCT Number)
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CHOEP + G-CSF followed by BEAM — CHOEP:
  Cyclophosphamide: 750 mg/m2 i.v. day1 Hydroxydaunorubicin: 50 mg/m2 i.v. day1 Vincristine: 1.4 mg/m2 (max 2 mg) i.v. day 1 Etoposide: 100 mg/m2 i.v. day 1-3 Prednisone: 100 mg daily p.o. day 1-5
  BEAM:
  Carmustine: 300 mg/m2 i.v. day 1 Etoposide: 100 mg/m2 i.v. x2 daily day 2-5 Cytosine arabinoside: 200 mg/m2 i.v. x2 daily or 400 mg/m2 as continuous 24 hrs i.v. infusion, day 2-5 Melphalan: 140 mg/m2 i.v. day 6

SUMMARY:
This is a phase II prospective non-randomised clinical trial in newly diagnosed and previously untreated adult patients in the age range 18-60 (67) years with peripheral T-cell lymphoma.

The treatment schedule will consist of three phases: induction and high-dose consolidation, followed by autologous stem cell rescue. There will be two different induction schedules: one for patients in the age range 18-60 years and one for patients aged over 60 years.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with newly diagnosed peripheral T-cell lymphoma of all stages. However, patients with nodal stage IA non-bulky disease (<10cm) can be treated individually at the discretion of the responsible physician.
* Following histologic subtypes (WHO classification) are eligible for inclusion in the study:

Peripheral T-cell lymphomas, unspecified Angioimmunoblastic T-cell lymphoma NK/T nasal-type T-cell lymphoma Enteropathy-type T-cell lymphoma Primary systemic, alk-negative anaplastic large cell lymphoma (T-or null phenotype) Hepatosplenic T-cell lymphoma Subcutaneous panniculitis-like T-cell lymphoma

NB: Patients should not enter the treatment program before confirmation of the histo-pathological diagnosis by the referral center pathologist

* Age 18-60 years. Patients in the age range 61-67 years may be included in this protocol at discretion of the treating physician.
* formed consent based on oral and written patient information (Appendix I)

Exclusion Criteria:

* Primary cutaneous T-or null-cell anaplastic large-cell lymphoma
* Alk-positive, primary systemic T-or null-cell anaplastic large-cell lymphoma
* WHO Performance Status grade 4 (Appendix II)
* Patients with severe cardiac (i.e. severe heart failure requiring symptomatic treatment or a cardiac ejection fraction of less than 45%), pulmonary, neurologic, psychiatric, renal, hepatic or metabolic disease.
* Pregnancy. N.B: Women of childbearing potential should be strongly advised to apply appropriate contraceptive precautions during the entire treatment period.
* Patients with concomitant malignancies except for non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Patients with seropositivity for the human immunodeficiency virus.
* Patients with other active and therapeutically uncontrolled infection.
* Psychological, familial, social or other condition/-s potentially hampering compliance and follow-up.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2001-10; Primary Completion 2008-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesco d'Amore, MD, Principal Investigator — Nordic Lymphoma Group
Locations (9):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Copenhagen Hospital, Copenhagen
  - Vejle Hospital, Vejle
- Finland (2):
  - OULO University Hospital, Oulu, Oulo
  - Kuopio University Hospital, Kuopio
- Norway (4):
  - Oslo University Hospital, Oslo
  - Ullevaal University Hospital, Oslo
  - Rogaland Hospital, Rogaland
  - St.Olavs Hospital, Trondheim